CLINICAL TRIAL: NCT06795789
Title: The Impact of a Multivitamin Combined Blueberry Polyphenol Supplement on Cognitive Function: A Pilot Study
Brief Title: Multivitamin Intervention and Cognitive Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Braincare Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Vitals_CF_01
Record Dates: First submitted 2025-01-09; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adult; Cognitive Measures
Keywords: Multivitamin; Polyphenols; Blueberry; Cognitive Function; Homocysteine; B-vitamins; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitals+ (combined multivitamin and polyphenol supplement) (Experimental): Participants to supplement with Vitals+ multivitamin combined polyphenol supplement for 3 months
  Interventions: Dietary Supplement: Vitals+ (combined multivitamin and polyphenol supplement)

INTERVENTIONS:
Dietary Supplement: Vitals+ (combined multivitamin and polyphenol supplement) — Multivitamin with 19 essential nutrients combined with Bilberry polyphenols
  Other Names: Vitals+

SUMMARY:
The purpose of this trial is to learn how a multivitamin combined blueberry polyphenol supplement (Vitals+) influences cognitive function in healthy adults. A secondary aim is to see how the biochemical level of nutritional factors change with the supplement.

This study will be completed fully remote (from the participants home without in-person visits). Participants will be asked to compete three steps over the course of 3 months:

Step 1:

Participants will be asked to complete an online cognitive function game (45 minutes)

Step 2:

Participants will receive a fingertip blood sample kit in the post to measure nutritional markers in the body (requiring 8 drops of blood). They will then be asked to complete the same online cognitive function game and answer some questions about their general health (50 minutes). After this, participants will be requested to start their multivitamin (Vitals+) subscription, once a day for 3 months.

Step 3:

This final step is the same as step 2. After 3 months participants will receive another fingertip blood sample kit in the post (requiring 8 drops of blood) and asked to complete the cognitive function games again (50 minutes). This will mark the end of the study.

How these measurements responded to the multivitamin supplement will then be measured.

DETAILED DESCRIPTION:
This study will investigate the influence of a 3 month multivitamin combined blueberry polyphenol supplement (Vitals+) on cognitive function, as measured by a validated online cognitive function test. The secondary outcome of this study is to evaluate nutritional biomarker response to the intervention. Specifically, elevated homocysteine concentrations have been reported as a risk factor for cognitive impairment and Dementia. Significant improvements in biomarker status of B-vitamins involved in homocysteine metabolism were found following intervention with this supplement (Vitals+). Therefore, it is hypothesised that the intervention will lead to reductions in homocysteine levels.

Furthermore, Vitamin D is a nutrient of concern, with deficient or suboptimal biomarker status reported across many European populations (particularly in winter months). Whilst vitamin D intervention has been shown to improve cognitive function in healthy adults. Therefore, a secondary hypothesis is that the supplement will lead to increased Vitamin D biomarker status.

It is hypothesised that any observed changes in cognitive function will be associated with changes in the biomarker response of homocysteine and Vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men and Women age >18 years
* Newly subscribed to the nutritional supplement
* Access to a PC or laptop with internet connection

Exclusion Criteria:

* Unable to give informed consent
* Consumed a nutritional supplement in past 3 months
* Consuming > 4 portions of B-vitamin fortified foods a week
* Pregnant or breastfeeding
* Diagnosis of a neurological condition, such as Dementia, depression or anxiety
* Prescribed vitamin B12 injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | 3 months
  A validated online Cognitive Function test will be used to assess cognition pre-post intervention

SECONDARY OUTCOMES:
Total homocysteine | 3 months
  Total homocysteine concentrations will be measured through blood spot samples by isotopic dilution and high-performance liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS)
Vitamin D | 3 months
  Vitamin D concentrations will be measured through blood spot samples by isotopic dilution and high-performance liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Harry R Jarrett, Ph.D, Principal Investigator — Heights
Locations (1):
- Heights Research and Development, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No